CLINICAL TRIAL: NCT05657067
Title: Effectiveness and Feasibility of Structured Emotionally Focused Family Therapy: A Pilot Study
Brief Title: Effectiveness and Feasibility of Structured EFFT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Principal Investigator, Henk Jan Conradi, PhD, Assistant Professor, University of Amsterdam
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-CP-15102; 2022-CP-15102 (Other: Ethics Review Board University of Amsterdam)
Record Dates: First submitted 2022-11-27; First posted 2022-12-20 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Emotion Regulation
Keywords: Attachment; Adolescents; Family; Mental Health Problems; Emotionally Focused Family Therapy (EFFT)
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emotionally Focused Family Therapy (EFFT) (Experimental): For this pilot study we aim for 15-20 included families who will be treated by three to five family therapists.
  Interventions: Behavioral: Emotionally Focused Family Therapy (EFFT)

INTERVENTIONS:
Behavioral: Emotionally Focused Family Therapy (EFFT) — The rationale behind EFFT is that mental health problems in children and adolescents often originate and/or are exacerbated by negative interaction patterns rooted in insecure attachment bonds within families. Therefore, the main treatment goal of EFFT is the development of secure attachment between parents and their children.

SUMMARY:
The goal of this clinical pilot study is to assess effectiveness and feasilibity of structured Emotionally Focused Family Therapy (EFFT) for parents and adolescents.

Participants will fill out questionnaires before, during and after the EFFT treatment Finally, feasibility will be assessed by semi-structured interviews.

DETAILED DESCRIPTION:
Background

The prevalence of mental health problems of children and adolescents worldwide is substantial with 10-20%. Attachment related emotion regulation is considered an important transdiagnostic process underlying mental health problems in adolescents. Emotionally Focused Family Therapy (EFFT) aims at the development of secure attachment between parents and their children in order to reduce the child's vulnerability for mental health problems and enhance resilience.

Intervention

The current pilot study is a first test of the newly developed protocol of structured EFFT. It consists of 4 phases and 16-21 sessions: phase 1 (1-2 sessions with the whole family) reframing the individual adolescent's problem as related to insecure attachment relations with the parents; phase 2A (4-6 sessions with the parents) and phase 2B (3 sessions with the adolescent) are delivered in parallel fashion and aim to prepare them to phase 3 by exploring insecure attachment relations and unfulfilled attachment needs; phase 3 (3 sessions with parents and adolescent) is focused on development of secure attachment relations between parents and adolescent; phase 4 (3 sessions with the whole family) consolidation of secure attachment and additional interventions for residual psychopathology; and finally a booster session with the whole family. Treatment adherence will be assessed with a check list by independent raters of sound recordings of random sessions.

Design and method

A within-subjects design, without randomized control group, with three waves will be applied: (1) waiting period of 2 months, (2) treatment phase 3-4 months, and (3) 2 months follow-up period concluded with a booster session. Comparing change during the waiting period vs. change during treatment will provide a clear indication of spontaneous remission vs. treatment-related change. The study will use a multi-method approach: quantitative for the effectiveness part (multilevel analyses of questionnaires) and qualitative for the feasibility part (semi-structured interviews). Treatment adherence will be assessed with sound recording of random sessions.

Hypotheses

Concerning the effectiveness of structured EFFT the researchers anticipate that, if limited power of this pilot study yields significant differences, outcomes will show:

1. no, or less change during the waiting period compared with the treatment phase;
2. gain during the treatment phase;
3. and substantial maintenance during follow-up. Hypotheses will be tested with multi-level analyses. Feasibility will be explored.

ELIGIBILITY:
Inclusion criteria:

For this pilot study we will include families with

1. adolescents aged 12-18 years (the so called 'identified' patient), and
2. families coping with mild problems.

Exclusion criteria:

The latter means that we will exclude:

1. blended families because of the more complex loyalties that exist between children and stepparents,
2. families of which individual members cope with serious trauma such as sexual and physical abuse and severe neglect, and
3. families of which the parents or children are diagnosed with severe DSM disorders (substance abuse or psychosis).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change from the waiting period in Negative interaction patterns on the Relationship Dynamics Scale (RDS; Stanley et al., 2001) during and after EFFT. | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The RDS is a validated self-reported 4 item questionnaire assessing negative interaction patterns over the past 2 weeks. Possible total scores range from 4 (negligible) to 16 (often). Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.
Change from the waiting period in Accessibility and responsiveness of the attachment figures on the Accessibility, Responsiveness, Emotional Engagement questionnaire (ARE; Johnson, 2008). | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The ARE is a validated self-reported 6 item questionnaire assessing accessibility and responsiveness of the attachment figures over the past month. Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.
Change from the waiting period in Discipline on the Discipline subscale of the Self-Efficacy for Parenting Tasks Index Toddler Scale (SEPTI; Coleman & Karraker, 2003). | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The Discipline 7 item subscale is part of the SEPTI a validated self-reported questionnaire assessing displine of the children by their partners over the past month. Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.
Change from the waiting period in Attachment between parents and adolescent and the parents as partners on the Experiences in Close Relationships - Relationship Structures questionnaire (ECR-RS; Fraley et al., 2011) | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The ECR is a validated self-reported 9 item questionnaire assessing Anxiety about rejection and abandonment and Avoidance of intimacy. Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.
Change from the waiting period in Relationship satisfaction between the parents as partners on the Couple Satisfaction Index (CSI; Funk & Rogge, 2007). | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The CSI is a validated self-reported 4 item questionnaire assessing relationship satisfaction over the past week. Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.
Change from the waiting period in the adolescent's Complaints on the Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997). | Through study completion, an average of 1 year per family: t1 = pre-waiting period; t2 = pre-treatment; t3 = pre-phase 3 (after 5-8 sessions); t4 = post treatment (after 16-21 sessions), t5 = pre-booster session (two months after final session)
  The SDQ is a validated self-reported 20 item questionnaire assessing adolescent's Complaints over the past month. Change will be assessed for: the waiting period (pre-treatment score - pre waiting period score), during EFFT (post treatment - pre treatment), during follow up (pre-booster session score - post -treatment score) and over the total study period.

SECONDARY OUTCOMES:
Feasibility of structured EFFT. | Two months after the final session, after the booster session has taken place. Semi-structured interviews will take place with the adolescent being interviewed separately from his or her parents.
  Feasibility will be assessed by semi-structured interviews.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychologiepraktijk Lenny Rodenbrug, Bussum, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data management The data will be saved under administration numbers to which each family member is linked and stored on the protected ICT environment of the University of Amsterdam. The data analysis will be performed at the University of Amsterdam. Personal data will be handled conform the General Data Protection Regulation.

REFERENCES:
- [Derived] Conradi HJ, Meuwese D, Rodenburg L, Dingemanse P, Mooren T. Effectiveness and feasibility of structured emotionally focused family therapy for parents and adolescents: Protocol of a within-subjects pilot study. PLoS One. 2023 Jun 23;18(6):e0287472. doi: 10.1371/journal.pone.0287472. eCollection 2023. PMID 37352284
- See also: This is the preregistration at the Open Science Framework which was published before recruitment commenced. The study protocol described at OSF is identical to the one provided here. — https://osf.io/39dt2/